CLINICAL TRIAL: NCT06628505
Title: Targeted Auditory Plasticity Training to Improve Central Hearing in Mild Traumatic Brain Injury (mTBI)
Brief Title: Auditory Plasticity Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000423; TP230338P1 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-08-29; First posted 2024-10-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Auditory plasticity; Hearing training
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial which will randomize subjects into one of two aims. Each aim will have a 1:1 randomization of participants into either the investigational or the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Speech in Noise Training (SPiN) (Active Comparator): Young to middle-age mTBI patients (age 18-55 yrs.) with various degrees of central hearing impairment will be randomly assigned to this training group
  Interventions: Other: Speech in Noise Training
- SPiN Control Group Treatment as Usual (TAU) (No Intervention): Young to middle-age mTBI patients (age 18-55 yrs.) with various degrees of central hearing impairment will be randomly assigned to a treatment as usual group
- Spatial Hearing Training (Active Comparator): Young to middle-age mTBI patients (age 18-55 yrs.) with various degrees of central hearing impairment will be randomly assigned to this training group
  Interventions: Other: Spatial Hearing Training Group
- Spatial Hearing Training Control Group Treatment as Usual (TAU) (Other): Young to middle-age mTBI patients (age 18-55 yrs.) with various degrees of central hearing impairment will be randomly assigned to a treatment as usual group
  Interventions: Other: Spatial Hearing Control Group

INTERVENTIONS:
Other: Speech in Noise Training — The active controls will receive frequency discrimination training that uses the same visual landscape and basic task of controlling the wisp based on judgments about acoustic cues. The task requires participants to avoid obstacles by swiping upward or downward on the touchscreen to indicate whether a test frequency associated with the obstacle was higher or lower, respectively, than a target sound presented slightly before the test sound.
  Other Names: SPiN
  Arms: Speech in Noise Training (SPiN)
Other: Spatial Hearing Training Group — Stimulus presentation and response measurement (Aim 2): Acoustic stimuli will be presented with a 360° speaker array that are fixed in place behind an opaque, nearly sound transparent, acoustic fabric curtain to avoid visual influences. Manual responses will be collected using a keyboard. Custom Matlab scripts control all relevant variables with millisecond precision. A webcam monitors the participant (not recorded) for the sole purpose of making sure the participant is always facing straight ahead.
  Sound localization task and training: Participants will judge the location of a target white noise sound (1000 ms, 70 dB SLP, 10-10,000 Hz) by moving an auditory pointer that appears 2 seconds after the offset of the target sound.
  The training group are given feedback about how their perceived location related to the actual sound location.
  Arms: Spatial Hearing Training
Other: Spatial Hearing Control Group — Stimulus presentation and response measurement (Aim 2): Acoustic stimuli will be presented with a 360° speaker array that are fixed in place behind an opaque, nearly sound transparent, acoustic fabric curtain to avoid visual influences. Manual responses will be collected using a keyboard. Custom Matlab scripts control all relevant variables with millisecond precision. A webcam monitors the participant (not recorded) for the sole purpose of making sure the participant is always facing straight ahead.
  Sound localization task and training: Participants will judge the location of a target white noise sound (1000 ms, 70 dB SLP, 10-10,000 Hz) by moving an auditory pointer that appears 2 seconds after the offset of the target sound.
  The training group are NOT given feedback about how their perceived location related to the actual sound location.
  Other Names: The training group performs the same spatial hearing task, but on every trial they are given feedback about how their perceived location related to the actual sound location.
  Arms: Spatial Hearing Training Control Group Treatment as Usual (TAU)

SUMMARY:
The investigators are working on a project to help people who have had mild brain injuries hear better. Sometimes, these injuries can make it hard for people to hear clearly, especially in noisy places or when trying to tell where sounds are coming from.

The project is testing special training exercises that have helped healthy people improve their hearing in these situations. The goal is to see if these exercises can also help people with mild traumatic brain injuries (mTBI).

If these exercises work, they could help doctors give better treatment to people with hearing problems after a brain injury. This would be especially helpful for soldiers who need to stay ready for duty. It could also make life better for veterans who struggle with hearing issues and help lower the cost of healthcare.

DETAILED DESCRIPTION:
The study has two aims:

1. Aim 1 - Speech in noise (SPiN) training: The training group will receive the SPiN training, while the active control group will play a variation of the main Listen game (frequency discrimination) that is not expected to improve speech recognition in noise. Participants will receive a tablet and earphones. The instructions will be explained, and they will practice and work with the experimenter to verify they understand how to run the training at home. Participants will do SPiN and Active Control training at home over 8 days, with up to two, 10 min sessions each day, for a total of 15 training sessions.
2. Aim 2 - Spacial hearing training: Two groups will be tested: training and control, and participants will be randomly assigned to one of two groups. The training group will receive Spatial Hearing training, which will be compared to no-contract controls. The study team will avoid withholding training from the controls by considering them a waitlist control group, which will then be offered the training after completing the study as a control participant.The training group does the same spatial hearing task on two days, but on every trial they are given feedback about how the location they thought the sound came from differed from the actual sound location.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* English is the primary language
* History of mTBI by self report

Exclusion Criteria:

* Pure tone threshold (mean of 0.5-4.0 kHz) > 40dB HL
* Major neurological or psychiatric conditions besides mTBI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Composite Hearing in Noise Score | Baseline to 1 month + 10 days
  The composite score will be the averaging (equal weighting) of z-scores from two tests: Spatial Release from Masking and Digits in Noise. Each test uses measures of decibels (dB), where smaller dB values indicate better performance.
Change in Frequency Following Response (FFR): Cross Correlation of FFR and Stimulus | Baseline to 1 month + 10days
  The time point of maximum correlation between the FFR and stimulus waveforms will be calculated. Larger correlation values indicate a more precise neural representation of the stimulus. A Fisher r-to-z transformation will be used to normalize the distribution of correlation values.
Change in Frequency Following Response : Amplitude of stimulus fundamental frequency | Time Frame: Baseline to 1 month + 10days
  The amplitude of the fundamental frequency will be defined using fast Fourier-transforms, and measured in microvolts. Larger values indicate greater amplitudes.
Change in Spatial Hearing: Sound localization Precision | Baseline to 1 month + 4 days
  Sound localization precision will be measured as the absolute difference (in degrees) between the locations of the pointer and the sound target location in the horizontal plane. Smaller values indicate better spatial hearing precision.
Change in Spatial Hearing: percent of front/back confusions. | Baseline to 1 month + 4 days
  Localization errors > 45° that cross the interaural axis will be categorized as front/back confusions. The percentage of Front/back confusions among all trials will be measured, and larger percentages indicate worse spatial hearing.
Change in P300 amplitude. | Baseline to 1 month + 4 days
  Amplitude of the P300 event-related potential in response to target sounds will be measured (in microvolts). Larger amplitudes indicate better spatial attention processing.

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Norman, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States